CLINICAL TRIAL: NCT03989219
Title: Methylation of cfDNA in Diagnosing and Monitoring Benign and Malignant Pulmonary Nodule
Brief Title: Methylation of cfDNA in Diagnosing and Monitoring Pulmonary Nodule
Status: Completed | Type: Observational
Sponsor: Jiayuan Sun (Other)
Responsible Party: Sponsor-Investigator, Jiayuan Sun, Chief Physician, Department of Pulmonary Medicine, Director, Department of Respiratory Endoscopy and Interventional Pulmonology, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Other Study IDs: SHCHE201802
Record Dates: First submitted 2019-06-16; First posted 2019-06-18 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Pulmonary Nodule, Solitary
Keywords: cfDNA methylation; CT follow-up; plasma; pulmonary nodule
MeSH Terms: conditions — Solitary Pulmonary Nodule

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Total cfDNA was extracted from 10ml plasma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- lung nodules were found by CT scanning: Plasma cfDNA will be performed in patients with pulmonary nodules (0.5-3 cm) found by CT scanning. Evaluation of benign and malignant diagnostic efficacy of cfDNA methylation in pulmonary nodules with clear pathological findings. Pulmonary nodules that could not or temporarily not require invasive examination will be performed CT follow-up and dynamically monitored methylation changes of cfDNA.
  Interventions: Procedure: plasma cfDNA methylation

INTERVENTIONS:
Procedure: plasma cfDNA methylation — plasma cfDNA will be performed in patients with pulmonary nodules (0.5-3 cm) found by CT scanning. Evaluation of benign and malignant diagnostic efficacy of cfDNA methylation in pulmonary nodules with clear pathological findings. Pulmonary nodules that could not or temporarily not require invasive examination will be performed CT follow-up and dynamically monitored methylation changes of cfDNA.

SUMMARY:
Patients found pulmonary nodules by CT screening by will be enrolled in this study prospectively. Plasma cfDNA sequencing of these patients will be used to diagnose and monitor benign and malignant pulmonary nodules.

DETAILED DESCRIPTION:
This study prospectively included patients with pulmonary nodules (0.5-3 cm) diagnosed by CT. Methylation of plasma cfDNA in these patients will be performed. Evaluation of benign and malignant diagnostic efficacy of cfDNA methylation in pulmonary nodules with definite pathological findings. Pulmonary nodules that temporarily not require invasive examination will be performed CT follow-up and dynamically monitored methylation changes of cfDNA. And the methylation changes were to establish a model for the diagnosis and monitor of benign and malignant pulmonary nodules.

ELIGIBILITY:
Inclusion Criteria:

* 1. Inclusion criteria:

  1. Aged 40-80;
  2. Lung nodules were detected by CT (≥5mm，≤3cm);
  3. Patients fully understand the informed consent and can sign the informed consent in person.

Exclusion Criteria:

* 2. Exclusion criteria:

  1. Patients diagnosed with malignant tumors in the past;
  2. This image suggests pulmonary nodules with hilar or mediastinal lymph node enlargement；
  3. Pulmonary nodules are suspected of intrapulmonary metastasis of lung cancer or other malignancies；
  4. Past diseases or conditions that affect plasma cfDNA content, such as rheumatoid immunity and diseases of the blood system.
  5. The researchers concluded that there were other conditions that made it inappropriate to participate in this study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of this study are those who meet the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
The efficacy of cfDNA methylation in the diagnosis of benign and malignant pulmonary nodules | 12 months
  The sensitivity, specificity, positive predictive value, negative predictive value and accuracy are calculated according to standard definitions to evaluate the efficacy of cfDNA methylation in the diagnosis of benign and malignant pulmonary nodules .

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, PhD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li Y, Xie F, Zheng Q, Zhang Y, Li W, Xu M, He Q, Li Y, Sun J. Non-invasive diagnosis of pulmonary nodules by circulating tumor DNA methylation: A prospective multicenter study. Lung Cancer. 2024 Sep;195:107930. doi: 10.1016/j.lungcan.2024.107930. Epub 2024 Aug 11. PMID 39146624